CLINICAL TRIAL: NCT04981288
Title: Lipids and Energy Study: Optimizing the Analysis of Lipids and Energy Metabolism in Blood Samples
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Martha Belury, Associate Professor, Ohio State University Comprehensive Cancer Center
Other Study IDs: 2021H0184
Record Dates: First submitted 2021-07-15; First posted 2021-07-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed research is a feasibility pilot trial designed to optimize the remote collection dried blood spots (DBS) from a finger stick and the analysis of fatty acid from the DBS and to optimize the analysis of mitochondria activity (or energy metabolism) from peripheral blood mononuclear cells (PBMC) or white blood cell samples. Participants in this study will provide a blood sample from venous blood draw and finger sticks. One finger stick collection will be completed remotely using a DBS kit that is sent through the mail while the other finger stick collection will be completed at the research site. These samples will be use to optimize the method for measuring fatty acids and mitochondria function as well as measure other lipids, insulin, glucose and markers of inflammation using established protocols. Demographic, dietary, sleep, and physical activity information will be measured using questionnaires, while height and weight will be measured to calculate body mass index (BMI).

DETAILED DESCRIPTION:
The primary objectives of the study are

* To optimize remote blood collection and laboratory analysis of polyunsaturated fatty acids (PUFAs) in dried blood spot (DBS) samples
* To optimize the analysis of mitochondria function in fresh and frozen peripheral blood mononuclear cells (PBMC)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Nonsmoking

Exclusion Criteria:

* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population chosen for the study is adults 18 years of age or older and strive to represent the ethnic diversity of the greater Columbus, OH region
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Optimize mitochondria function measurements in fresh and frozen blood | 1 Day
  Measuring oxygen consumption rate in peripheral blood mononuclear cells using seahorse analyzer
Optimize remote blood collection and laboratory analysis of in dried blood spot samples | 2 Days
  Collecting dried blot spots remotely and in the research setting and venous blood draw in the research setting to compare fatty acid composition

SECONDARY OUTCOMES:
Assess the relationship of mitochondria function in and cardiolipin in peripheral blood mononuclear cells | 1 Day
  Determine mitochondria function in peripheral blood mononuclear cells by measuring oxygen consumption rate and determining its relationship to the mitochondrial phospholipid cardiolipin
Assess the relationship of mitochondria function and fatty acid metabolites | 1 Day
  Determine mitochondria function in peripheral blood mononuclear cells by measuring oxygen consumption rate and determining its relationship to the fatty acid metabolites in plasma
Assess the relationship of mitochondria function and markers of inflammation | 1 Day
  Determine mitochondria function in peripheral blood mononuclear cells by measuring oxygen consumption rate and determining its relationship to markers of inflammation in plasma
Assess the relationship of mitochondria function in peripheral blood mononuclear cells and markers of glycemia | 1 Day
  Determine mitochondria function in peripheral blood mononuclear cells by measuring oxygen consumption rate and determining its relationship to markers of glycemia in serum

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Human Nutrition Laboratory, Columbus, Ohio, United States